CLINICAL TRIAL: NCT01110213
Title: Goal Setting and Decisional Balance Applied to Physical Activity and Fruit & Vegetable Consumption
Brief Title: Goal Setting and Lifestyle
Acronym: GSDB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Collaborators: University of Hawaii Cancer Research Center (Other)
Responsible Party: Raheem Paxton, Postdoctoral Fellow, University of Texas M D Anderson Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHS - 14544
Record Dates: First submitted 2010-04-21; First posted 2010-04-26 (Estimated); Last update posted 2010-04-26 (Estimated); Status verified 2010-04

CONDITIONS: Physical Activity; Diet
Keywords: Aging; physical activity; diet; goal setting
MeSH Terms: conditions — Motor Activity | interventions — Exercise; Fruit; Vegetables

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physical activity (Experimental): Participants received individual tailored telephone counseling and group-tailored newsletters encouraging leisure time physical activity. Content was based on goal setting theory and decisional balance.
  Interventions: Behavioral: Physical activity
- Fruit and vegetable (Experimental): Participants received individual tailored telephone counseling and group-tailored newsletters encouraging fruit and vegetable intake. Content was based on goal setting theory and decisional balance.
  Interventions: Behavioral: Fruit and vegetable

INTERVENTIONS:
Behavioral: Physical activity — Participants received two individually tailored phone calls and two condition specific newsletters encouraging goal setting and weighing the pros and cons for physical activity.
  Arms: Physical activity
Behavioral: Fruit and vegetable — Participants received two individually tailored phone calls and two condition specific newsletters encouraging goal setting and weighing the pros and cons for fruit and vegetable consumption.
  Arms: Fruit and vegetable

SUMMARY:
The primary aim of this feasibility study is to determine if a theory-based lifestyle intervention consisting of telephone counseling is associated with improvements in physical activity and dietary intake.

DETAILED DESCRIPTION:
Goal setting has become an integral part of physical activity and dietary interventions; however, few studies have examined the theoretical constructs that drive goal-setting theory. To address the limitations and gaps in the literature, we designed an 8-week health behavior intervention for a racially and ethnically diverse sample of older adults. The primary aim of this study was to determine whether older adults randomized to a goal-setting intervention for physical activity or fruit and vegetable (F&V) intake would make significant improvements in physical activity or F&V intake. The secondary aim of this study was to determine whether participating in goal-setting interventions was associated with changes in theoretical constructs related to goal-setting. We hypothesized that older adults assigned to the physical activity condition would significantly increase metabolic minutes (MET-minutes) of physical activity from baseline to follow-up and that participants assigned to the F&V intake condition would significantly increase mean servings of F&V. In addition, we hypothesized that mean scores of goal specificity, difficulty, effort, commitment, persistence, barrier self-efficacy, and task self-efficacy would significantly increase from baseline to follow-up for both groups.

ELIGIBILITY:
Inclusion Criteria:

* must be 55 years or older,
* posses a telephone,
* able to give informed consent, and
* commit to a 10 week study.

Exclusion Criteria:

* currently enrolled in a study promoting physical activity or dietary intake,
* currently exceeding current recommendations for physical activity or F&V intake at baseline, and
* medical conditions contraindicating physical activity or fruit and vegetable consumption.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2006-08; Primary Completion 2007-03 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Leisure Time Physical Activity | 8-weeks
  Physical Activity was measured using an adaptation of the Godin Leisure-Time Exercise Questionnaire. Participants reported how many times during an average week they participated in mild (i.e., takes minimal effort), moderate (i.e., increases your heart and breathing rate a little), and strenuous activity (i.e., caused one's heart to beat rapidly) for at least 30 minutes at a time.

SECONDARY OUTCOMES:
Goal specificity and difficulty | 8-weeks
  Goal Specificity and Difficulty. Four items were created for each concept: (1) "The goals I set for number times I will [eat F&V or exercise] in a week are," (2) "the goals I set for the type of [F&V or exercise] I will [eat or do] in a week are," (3) "the goals I set for the [amount or duration] of [F&V or exercise] I get in a week are," and (4) "the goals I set for intensity of my exercise sessions within a week are."

CONTACTS AND LOCATIONS:
Overall Officials: Raheem J Paxton, PhD, Principal Investigator — University of Hawaii Cancer Research Center
Locations (1):
- Cancer Research Center of Hawaii / University of Hawaii, Honolulu, Hawaii, United States